CLINICAL TRIAL: NCT05708170
Title: Impact of Intravenous Iron (Ferinject) on Musculoskeletal Function Profiles in Older Adults With Iron Deficiency Anaemia (IDA)
Brief Title: Impact of Intravenous Iron on Musculoskeletal Function in Older Adults
Acronym: FERIDA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Liverpool Hope University (Other)
Collaborators: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: LHU-FERIDA
Record Dates: First submitted 2022-10-17; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-08

CONDITIONS: Iron Deficiency Anemia
Keywords: Iron Deficiency Anaemia; Skeletal Muscle Function; Musculoskeletal; Ageing
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; ferrous sulfate; Iron

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous iron therapy group (Experimental): This group will receive intravenous iron calculated based on body weight and level of anaemia (hemoglobin concentration), as per the iron therapy's SPC.
  Interventions: Drug: Ferinject
- Active Control Group (Active Comparator): This group will receive oral ferrous sulphate prescribed by their GP Randmisation: Simple randomisation/parallel assignment/single-blinded
  Interventions: Drug: Ferrous Sulfate 200 MG

INTERVENTIONS:
Drug: Ferinject — Ferinject Therapy Group: each patient's Iron need for repletion by the Ferinject will be determined using product SPC dosing based on patient's body weight and Hb level. Accordingly, the appropriate dose of Ferinject will be administered while ensuring that a single administration will not exceed:
  * 15 mg iron/kg body weight (for administration by intravenous injection) or 20 mg iron/kg body weight (for administration by intravenous infusion)
  * 1,000 mg of iron (20 mL Ferinject) The cumulative dose of Ferinject per week will not exceed 1,000 mg of iron (20 mL Ferinject).
  Other Names: ferric carboxymaltose
  Arms: Intravenous iron therapy group
Drug: Ferrous Sulfate 200 MG — Active Control Group (standard care excl. IV Iron): Oral Ferrous sulphate 200 mg three times daily.
  Other Names: oral iron
  Arms: Active Control Group

SUMMARY:
Anaemia is a risk factor for functional decline and frailty in older adults including decreased physical performance and muscle strength, increased hospitalisation risk and mortality, falls, and poorer recovery from activities of daily living. Despite a major gap in human studies, research in animals has demonstrated an interrelationship between iron deficiency anaemia and deteriorated functional capacity and physical performance particularly in older adults. Iron deficiency and associated anaemia is a frequent accompanier of debilitating chronic diseases such as heart failure and chronic lung diseases. These conditions, more commonly seen in older patients, are strongly linked to deterioration in physical function, reduced skeletal muscle mass and quality, frailty, and poor quality of life. Exercise intolerance is also a common feature of these conditions as iron deficiency impairs the capacity of carrying oxygen leading to inability to sustain physical activities. Furthermore, the age-related decline in the muscle mass and quality (so called sarcopenia) and associated frailty has rapidly become a major health concern in the older adults particularly when accompanied by other chronic diseases. Recently, there has been an increasing interest in exploring the role of iron as a causative factor in the development of sarcopenia and related frailty.

In summary, there is a substantial gap of evidence whether Iron repletion leads to meaningful enhancements in the skeletal muscle function and physical performance in older adults suffering from iron deficiency anaemia. This study will investigate the impact of a standard care intervention (intravenous iron therapy) on muscular function and physical performance in older patients through a range of laboratory assessments.

DETAILED DESCRIPTION:
The study will recruit two groups of stable patients (although likely with chronic diseases) with established iron deficiency anaemia through Aintree Hospital NHS Trust clinics. Fifty patients aged 60-85 years will be recruited into each group:

1. Intravenous iron therapy group: This group will receive intravenous iron calculated based on body weight and level of anaemia (hemoglobin concentration), as per the iron therapy's SPC
2. Active Control Group: This group will receive oral ferrous sulphate prescribed by their GP Randmisation: Simple randomisation/parallel assignment/single-blinded

Identified patients with iron deficiency anaemia will receive an invitation to participate in the study together with a Patient Information Sheet clearly explaining different aspects of the research project. Each participant will require to attend the School of Health Sciences' laboratories (Liverpool Hope University) on four different occasions (once before the intervention and three times after receiving the iron therapy) throughout a 3-year period to complete multiple assessments in relation to basic blood tests and musculoskeletal function and physical performance. In addition to this, participants in the first group will require to attend the Aintree Hospital NHS Trust clinics on one occasion to receive a single-dose intravenous iron.

The study will broadly investigate musculoskeletal function (health) and physical performance by means of muscle quality, muscle mass, muscle strength, muscle activation and fatigue levels, gait quality, muscle physiology (level of oxygen carried into the muscles), and functional questionnaires prior to, during, and after iron therapy. In addition to this, changes in patients' quality of life in each group will be assessed through administration of validated questionnaires.

The data will be analysed at the end of the study to identify any significant and clinically meaningful changes in the musculoskeletal function, physical performance, and health-related quality of life resulted from the iron therapy in each group while also comparing such changes between the two study groups.

ELIGIBILITY:
Inclusion Criteria:

* Anaemia attributable to iron deficiency
* Haemoglobin < 120 g/L in women, Hb < 130 g/L in men
* Ferritin ≤100 ng/mL or ≤300 ng/mL if transferrin saturation (TSAT) ≤30%
* Age ≥ 60 to 85 years
* Ambulatory individuals
* Written informed consent

Exclusion Criteria:

* Patients already taking intravenous or oral iron
* BMI > 40 kg/m²
* Uncontrolled hypertension/ diabetes
* Potential medication interactions
* Hemochromatosis or iron storage disorders
* Recent treatment with IV antibiotics or red blood cell transfusion
* Dialysis dependent
* History of malignancy
* Pregnant or lactating women
* Severe hepatic and renal dysfunction
* Advanced cardiovascular disease and COPD
* Advanced Neuromuscular disorder
* Obvious cognitive disability and psychological illness
* Current treatment with systemic steroids or any other substantive medication
* Alcohol or any other drug abuse

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Muscle Quality Index (MQI) | "through study completion, an average of 2 year"
  Muscle strength relative to volume of the muscle mass generating the force

SECONDARY OUTCOMES:
Health-history Questionnaire | Baseline
  Questionnaire to document participant health history
International Physical Activity Questionnaire-IPAQ) | Baseline
  Questionnaire to determine the level of physical activity
Blood Iron Profile | "Through study completion, an average of 2 year"
  Blood analysis including Hemoglobin, Iron, Ferritin, and Transferrin
Upper Extremity Strength (in Newtons) | "Through study completion, an average of 2 year"
  Dynamometry to measure upper extremity (Grip and shoulder forward flexion) strength
Lower Extremity Muscle Strength (in Newtons) | "Through study completion, an average of 2 year"
  Dynamometry to measure lower extremity (Knee extension) strength
Skeletal Muscle Mass (kg) | "Through study completion, an average of 2 year"
  Bio-Impedance (BIA) to measure the skeletal muscle mass (kg)
Muscle Fatigue | "Through study completion, an average of 2 year"
  Electromyographic (EMG) assessment of localised muscle fatigue
Muscle Activation | "through study completion, an average of 2 year"
  Electromyographic (EMG) assessment of muscle activity level
Gait Analysis | "Through study completion, an average of 2 year"
  3-Dimensional Motion Capture to assess gait quality
Short Battery of Physical Performance (SBPP) | "through study completion, an average of 2 year"
  A validated test for assessing physcial and functional capacity
Mitochondrial Function | "through study completion, an average of 2 year"
  Near-infrared spectroscopy (NIRS) to investigate quality of oxidation in muscles
The 12-Item Short Form Health Survey (SF-12) | "Through study completion, an average of 2 year"
  A patient-rated questionnaire to assess the Quality of Life
The Hospital Anxiety and Depression Scale (HADS) | "Through study completion, an average of 2 year"
  A patient-rated questionnaire to assess anxiety and Depression
The Sarcopenia Quality of Life (SarQoL) | "through study completion, an average of 2 year"
  A patient-rated questionnaire to assess Sarcopenia-specific quality of life
The Upper Extremity Functional Index (UEFI) | "through study completion, an average of 2 year"
  A patient-rated questionnaire to assess Upper Extremity Function
The Lower Extremity Functional Index (UEFI) | "through study completion, an average of 2 year"
  A patient-rated questionnaire to assess Lower Extremity Function

IPD SHARING:
Plan to Share IPD: Undecided
NK

REFERENCES:
- See also: ISRCTN — https://www.isrctn.com/ISRCTN13325706
- See also: NHS/HRA — https://www.hra.nhs.uk/planning-and-improving-research/application-summaries/research-summaries/impact-of-intravenous-iron-on-musculoskeletal-function-in-older-adults/
- See also: WHO - International Trial Registry Platform — https://trialsearch.who.int/Trial2.aspx?TrialID=ISRCTN13325706